CLINICAL TRIAL: NCT04848142
Title: Psychosocial Impact of Disclosing Cancer Predisposition Genetic Testing Results During Childhood
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PSYGEN
Record Dates: First submitted 2021-04-12; First posted 2021-04-19 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Pediatric Cancer; Predisposition, Genetic
MeSH Terms: conditions — Neoplasms; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary Group (parent-child): parents (i.e., guardians/caregivers) and children age ≥ 8 years,will complete questionnaires to examine the impact of germline variant disclosure on parent adjustment, parenting, and child adjustment. Optional qualitative interviews may be completed individually for participants (age ≥ 12 years with P/LP variant and aware of results, or their parent)
- Parent Only Group: parents of children age < 8 years, will complete questionnaires to examine the impact of germline variant disclosure on parent adjustment, parenting, and child adjustment.

SUMMARY:
The participants are being asked to take part in this research study because the participant is a child who has been diagnosed with cancer and has completed genetic testing to find out if the participant has a variant in a gene that may predispose the participant to cancer, and/or the participants are the parents (i.e., guardian/caregiver) of this child. This research is being done to understand how finding out the results of genetic testing during childhood impacts the participant and family. The investigator will compare the emotions and behavior of parents and children based on the genetic testing results.

Primary Objective

* Examine the impact of genetic testing result disclosure for a pathogenic (P)/likely pathogenic (LP) germline variant in a known cancer predisposing gene versus negative results on parent adjustment (i.e., emotional functioning, cancer worry, symptom interpretation, and genetic testing related worry/distress).
* Examine the impact of genetic testing result disclosure for a P/LP germline variant versus negative results on parenting (i.e., responses to children's symptoms, overprotectiveness, parent-child communication, cohesion, and expressivity in the family).

Exploratory Objectives

* Examine the impact of genetic testing result disclosure (P/LP versus negative results) on child adjustment (i.e. emotional functioning, cancer worry, self-perception, and life meaning and purpose).
* Examine the impact of disclosing a variant of uncertain significance (VUS) on parent adjustment, parenting, and child adjustment.
* Examine the indirect association between genetic testing result disclosure (P/LP versus negative results) and child adjustment through parental adjustment and parenting behavior.
* Qualitatively identify children and parents' perspectives of how disclosure of a cancer predisposition has affected children's emotional, social, personal, and familial functioning.

DETAILED DESCRIPTION:
A mixed methods approach, including questionnaires and qualitative interviews with children and their parents. Participants ("Primary Strata:" parents (i.e., guardians/caregivers) and children age ≥ 8 years, n=132; "Parent Only Strata:" parents of children age < 8 years, n=66) will complete questionnaires to examine the impact of germline variant disclosure on parent adjustment, parenting, and child adjustment. Optional qualitative interviews may be completed individually for participants (age ≥ 12 years, n=30) with P/LP variants (and who are aware of their result status) and their parents (n=30) to obtain more open-ended information about the impact of genetic testing result disclosure, family communication about testing results, and their perception of result implications.

ELIGIBILITY:
Inclusion Criteria:

Primary Strata

* Patient underwent germline genetic testing as offered through the SJCRH Cancer Predisposition Program with results disclosed to patient and/or parents (i.e., of testing results are not a criterion for eligibility)
* Patient's age at the time of initial germline result disclosure was birth - 17 years of age (inclusive)
* Patient had diagnosis of malignancy (or benign tumor; e.g., craniopharyngioma) prior to germline testing
* A parent/legal guardian/caregiver is willing to participate in the research study and provide consent
* Participant family is fluent in English for completion of questionnaires (able to speak and read)
* Patient is currently 8 years of age or older

Parent Only Strata

* Parent (i.e., guardian/caregiver) of a patient who underwent germline genetic testing as offered through the SJCRH Cancer Predisposition Program with results disclosed to patient and/or parents 1 - 3 years (inclusive) previously (Note- patient's knowledge of testing results are not a criterion for eligibility)
* Parent of a patient whose age at the time of initial germline result disclosure was birth - 17 years of age (inclusive)
* Parent of a patient with a diagnosis of malignancy (or benign tumor; e.g., craniopharyngioma) prior to germline testing
* Parent/caregiver is a legal guardian willing to participate in the research study and provide consent
* Participant family is fluent in English for completion of questionnaires (able to speak and read).
* Parent of a patient currently younger than 8 years of age.

Exclusion Criteria:

* Inability or unwillingness of research participant or parent (i.e., guardian/caregiver) to give informed consent
* Parent is under the age of 18 years
* Parent has evidence of significant cognitive deficits (per medical report) that would interfere with the ability to comprehend questionnaires
* Research participant's medical status or condition precludes completion of the study (as determined by the medical team, patient, or parent)

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All participants who meet eligibility criteria and consent to enrollment on the study.
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2023-10-13 (Actual)

PRIMARY OUTCOMES:
Fear of Cancer Recurrence | Day 0
  Independent two-sample t-tests will assess statistical parental adjustment differences between group means (i.e., parents of children with pathologic/likely pathologic vs. negative genetic testing result) on the parent-reported Fear of Cancer Recurrence - Short Form. Only in the situation of outliers, two-sample Mann-Whitney U tests will be used for testing purposes.
Cancer Information Questionnaire for Parents | Day 0
  Independent two-sample t-tests will assess statistical parental adjustment differences between group means (i.e., parents of children with pathologic/likely pathologic vs. negative genetic testing result) on the Cancer Information Questionnaire for Parents. Only in the situation of outliers, two-sample Mann-Whitney U tests will be used for testing purposes.
Multidimensional Impact of Cancer Risk Assessment | Day 0
  Independent two-sample t-tests will assess statistical parental adjustment differences between group means (i.e., parents of children with pathologic/likely pathologic vs. negative genetic testing result) on the parent-reported Multidimensional Impact of Cancer Risk Assessment. Only in the situation of outliers, two-sample Mann-Whitney U tests will be used for testing purposes.
Brief Symptom Inventory 18 | Day 0
  Independent two-sample t-tests will assess statistical parental adjustment differences between group means (i.e., parents of children with pathologic/likely pathologic vs. negative genetic testing result) on the parent-reported Brief Symptom Inventory 18. Only in the situation of outliers, two-sample Mann-Whitney U tests will be used for testing purposes.
Impact of Event Scale | Day 0
  Independent two-sample t-tests will assess statistical parental adjustment differences between group means (i.e., parents of children with pathologic/likely pathologic vs. negative genetic testing result) on the parent-reported Impact of Event Scale - Revised. Only in the situation of outliers, two-sample Mann-Whitney U tests will be used for testing purposes.
Psychological Adaptation to Genetic Information Scale | Day 0
  Independent two-sample t-tests will assess statistical parental adjustment differences between group means (i.e., parents of children with pathologic/likely pathologic vs. negative genetic testing result) on the parent-reported Psychological Adaptation to Genetic Information Scale-Modified. Only in the situation of outliers, two-sample Mann-Whitney U tests will be used for testing purposes.
Symptom Interpretation Questionnaire-Parent Report | Day 0
  Independent two-sample t-tests will assess statistical parental adjustment differences between group means (i.e., parents of children with pathologic/likely pathologic vs. negative genetic testing result) on the Symptom Interpretation Questionnaire-Parent Report. Only in the situation of outliers, two-sample Mann-Whitney U tests will be used for testing purposes.
Parent-Adolescent Communication Scale | Day 0
  Independent two-sample t-tests will assess statistical parenting differences between group means (i.e., parents of children with pathologic/likely pathologic vs. negative genetic testing result) of parent- and child-reports on the Parent-Adolescent Communication Scale. Only in the situation of outliers, two-sample Mann-Whitney U tests will be used for testing purposes.
Family Environment Scale | Day 0
  Independent two-sample t-tests will assess statistical parenting differences between group means (i.e., parents of children with pathologic/likely pathologic vs. negative genetic testing result) on the parent-reported Family Environment Scale-Revised. Only in the situation of outliers, two-sample Mann-Whitney U tests will be used for testing purposes.
Parental Bonding Instrument | Day 0
  Independent two-sample t-tests will assess statistical parenting differences between group means (i.e., parents of children with pathologic/likely pathologic vs. negative genetic testing result) on the child-reported Parental Bonding Instrument. Only in the situation of outliers, two-sample Mann-Whitney U tests will be used for testing purposes.
Parent Protection Scale | Day 0
  Independent two-sample t-tests will assess statistical parenting differences between group means (i.e., parents of children with pathologic/likely pathologic vs. negative genetic testing result) on the parent-reported Parent Protection Scale. Only in the situation of outliers, two-sample Mann-Whitney U tests will be used for testing purposes.
Openness to Discuss Cancer in the Family | Day 0
  Independent two-sample t-tests will assess statistical parenting differences between group means (i.e., parents of children with pathologic/likely pathologic vs. negative genetic testing result) on the parent-reported Openness to Discuss Cancer in the Family. Only in the situation of outliers, two-sample Mann-Whitney U tests will be used for testing purposes.
Child Vulnerability Scale | Day 0
  Independent two-sample t-tests will assess statistical parenting differences between group means (i.e., parents of children with pathologic/likely pathologic vs. negative genetic testing result) on the parent-reported Child Vulnerability Scale. Only in the situation of outliers, two-sample Mann-Whitney U tests will be used for testing purposes.
Adult Responses to Children's Symptoms | Day 0
  Independent two-sample t-tests will assess statistical parenting differences between group means (i.e., parents of children with pathologic/likely pathologic vs. negative genetic testing result) on the parent-reported Adult Responses to Children's Symptoms. Only in the situation of outliers, two-sample Mann-Whitney U tests will be used for testing purposes.

CONTACTS AND LOCATIONS:
Overall Officials: Katianne Sharp, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St.Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St.Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols